CLINICAL TRIAL: NCT07008677
Title: Oral Health Awareness and Oral Health Status Among Professional Musicians in German Orchestras: An Online-Based Survey Study
Brief Title: Oral Health Awareness and Status Among Professional Musicians in German Orchestras
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Felix Marschner, Main Investigator, University Medical Center Goettingen
Other Study IDs: 2/5/25
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Oral Hygiene, Oral Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- German professional musicians: Professional orchestra musicians in Germany
  Interventions: Other: online questionaire

INTERVENTIONS:
Other: online questionaire — The online questionnaire includes demographic data: age, gender, instrument, professional background, and oral health behavior

SUMMARY:
Germany has the highest density of professional orchestras worldwide, comprising over 9,900 musicians in 129 ensembles. These musicians are exposed to specific occupational stressors that may impact not only their mental and physical well-being but also their oral health. The demands of rehearsals, performances, and long hours of instrument practice place unique strain on the body. In particular, wind instrument players are at an elevated risk of developing dental malocclusions and temporomandibular joint (TMJ) disorders due to prolonged and asymmetric pressure on the oral and facial structures. Such profession-related burdens may lead to a higher level of oral health awareness and a greater motivation to engage in preventive measures. Despite these factors, there is a lack of empirical data on the oral health awareness, oral health status, and preventive behavior of professional musicians. To date, no studies have systematically assessed these aspects within this occupational group, nor have differences between instrumental groups-such as woodwinds, brass, strings, percussion, or others like piano, harp, or celesta-been adequately explored.

The aim of this pilot study is to evaluate the level of oral health awareness and the willingness to engage in preventive behaviors among professional musicians in German orchestras. The study is conducted as a purely data-based, prospective, non-interventional online survey. It does not involve any clinical examinations, diagnostics, or therapeutic interventions. Instead, a standardized online questionnaire is used to collect data on demographic characteristics, professional background, and oral health behavior. The survey also includes questions on potential risk factors and the frequency of preventive dental care utilization. Participation is voluntary and anonymous. The only study-related activity is the one-time completion of the online questionnaire, which is not part of any clinical routine. The estimated time required to complete the questionnaire is approximately 10 minutes.

The study is exploratory in nature and is intended to generate baseline data that can serve as the foundation for future research and the development of targeted oral health prevention strategies tailored to the needs of musicians. Since this is a pilot study, no formal sample size calculation will be conducted. All professional musicians from the 129 German orchestras who meet the inclusion criteria-being at least 18 years old and working as professional musicians in either freelance or employed settings-will be invited to participate. The final sample size will be determined by the number of valid responses. Individuals who do not provide informed consent will be excluded from the study.

The primary outcomes of the study include the assessment of oral health awareness, identification of patterns in preventive behavior, and the analysis of potential differences between instrumental groups. In the long term, the results may help to highlight specific occupational health risks related to oral health in musicians and may inform the development of targeted prevention strategies and education programs. By collecting these data, the study contributes to filling a significant research gap and provides a foundation for improving the oral health and well-being of professional musicians.

ELIGIBILITY:
Inclusion Criteria:

* Musicians in professional German orchestras working freelance and/or under employment

Exclusion Criteria: co

* consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Musicians in professional German orchestras working freelance and/or under employment
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Online-questionaire | 10 minutes
  Completion of a web based questionnaire with demographic data

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided